CLINICAL TRIAL: NCT01442805
Title: Etude contrôlée Des Effets de la réalité Virtuelle Sur Les symptômes et Les paramètres Physiologiques de Certaines Phobies spécifiques
Brief Title: Use of Virtual Reality in the Treatment of Flying Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080102
Record Dates: First submitted 2011-09-15; First posted 2011-09-29 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Flying Phobia
Keywords: Cognitive Behavior Therapy; Virtual Reality Exposure Therapy; Psychophysiological Measures; Driving Phobia; Flying Phobia
MeSH Terms: conditions — Aerophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RV (Experimental): Cognitive Behavioral Therapy with Virtual Reality Exposures
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- IMAGO (Experimental): Cognitive Behavioral Therapy with Exposure Therapy through Imagination
  Interventions: Behavioral: Exposure Therapy through Imagination

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Participants are exposed to the feared situation (flying) through the virtual reality technology
  Arms: RV
Behavioral: Exposure Therapy through Imagination — Participants are exposed to the feared situation (flying) through exposure technique of imagination.
  Arms: IMAGO

SUMMARY:
The project aims to explore the potential of Virtual Reality Exposure Therapy (VRET) for the treatment of the fear of driving, the fear of flying and the fear of public speaking.

The study is a randomized controlled trial (RCT) designed to compare the efficiency of cognitive behavioural therapy with exposures in imagination to behavioural therapy with exposures in virtual reality. Anxiety levels are measured using specific questionnaires, SUD ratings and physiological measures (heart rate, skin conductance, skin temperature, breathing frequency, heart rate variability).

Hypothesis: Treatments with exposures in virtual reality are more efficient than treatments with exposures in imagination.

DETAILED DESCRIPTION:
In the past, several studies have demonstrated the effectiveness of virtual reality exposure therapy in the treatment of flying phobia and driving phobia. As an objective tool, psychophysiological recordings help demonstrate the decrease of physiological aspects of anxiety reactions (heart rate, skin conductance, skin temperature, heart rate variability and breathing pattern).

The aim of the present study is to examine the effects of cognitive behavioural therapy with exposures in imagination to behavioural therapy with exposures in virtual reality in the treatment of patients with flying phobia. Thirty patients will be randomized into either an imagination exposure group or a virtual reality exposure group after having received four sessions of cognitive behavioural therapy for coping with panic attacks. Respective exposure therapies consist in four sessions.

Anxiety levels will be measured before and after the cognitive behavioural therapy for coping with panic attacks as well as before and after the exposure therapy sessions and after 3 months using specific questionnaires, SUD ratings and psychophysiological measures (heart rate, skin conductance, skin temperature, breathing frequency and heart rate variability). The exposure stimuli will consist in a 10min movie of a flight with an insight-cabin viewing perspective.

The investigators hypothesize that virtual reality exposure therapies will be more effective than imagination exposure therapy in terms of decrease of anxiety self-ratings and psychophysiological fear reactions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a specific phobia (DSM-IV-TR)

Exclusion Criteria:

* Pregnant women
* Subjects with severe pulmonary / cardiovascular problems; Asthma, epilepsy, vertigo
* Drug abuse
* Subjects under on-stabilized anti-depressant treatment
* Psychotic subjects
* Subjects with suicidal ideas
* Subjects presenting insufficient intellectual capabilities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Flight taken | 6 months
  Participants are expected to take a real flight

SECONDARY OUTCOMES:
Physiological Measures | 6 months
  Heart Rate, Breathing frequency, Skin conductance, Skin Temperature, Heart Rate Variability
Specific Questionnaires | 6 months
  Specific Questionnaires: SUD, Motivational Scale, Fear Questionnaire Marks 1979, Sheehan Disability Scale, STAI I & II, BDI, BAI, GAF, Flight Anxiety Situations Questionnaire FAS, Flight Anxiety Modality Questionnaire FAM

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pull, Prof.Dr., Principal Investigator — Centre de Recherche Public de la Santé
Locations (1):
- Centre de Recherche Public de la Santé, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No